CLINICAL TRIAL: NCT06674954
Title: Comparison of Perioperative Characteristics of Regional Anasthesia and General Anesthesia in Shoulder Arthroscopy
Brief Title: Comparison of Perioperative Characteristics of Regional Anasthesia and General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Atakan Sezgi, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0125
Record Dates: First submitted 2024-10-16; First posted 2024-11-05 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Arthroscopy; Peripheral Nerve Block
Keywords: Shoulder Arthroscopy; General Anesthesia; Regional Anesthesia
MeSH Terms: interventions — Anesthesia, Conduction; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional anesthesia (Active Comparator): After the patients are monitored and in the supine position, after appropriate field sterilization, interscalene brachial plexus block, superficial cervical block, and supraclavicular brachial plexus block will be applied to these patients under ultrasound guidance. Total of 40 ml of local anesthetic solution (20 ml %0.5 bupivacaine + 10 ml %2 lidocaine + 10 ml physiological saline) will be prepared; 15 ml will be used for interscalene brachial plexus block, 10 ml will be used for superficial cervical block, and 15 ml will be used for supraclavicular brachial plexus block.
  Interventions: Procedure: Regional Anesthesia
- General anesthesia (Active Comparator): Anesthesia induction will be performed with 2.5 mg/kg propofol, 0.6 mg/kg rocuronium, and 1 mcg/kg fentanyl. Maintenance will be achieved with sevoflurane (MAC: 0.9-1.0) and remifentanil (0.05-0.2 mcg/kg/min). Remifentanil titration will be done according to basal heart rate and blood pressure.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Regional Anesthesia — After the patients are monitored and in the supine position, after appropriate field sterilization, interscalene brachial plexus block, superficial cervical block, and supraclavicular brachial plexus block will be applied to these patients under ultrasound guidance. Total of 40 ml of local anesthetic solution (20 ml %0.5 bupivacaine + 10 ml %2 lidocaine + 10 ml physiological saline) will be prepared; 15 ml will be used for interscalene brachial plexus block, 10 ml will be used for superficial cervical block, and 15 ml will be used for supraclavicular brachial plexus block.
  Tramadol (100 mg, intravenous) and dexketoprofen (50 mg, intravenous) will be administered intraoperatively as standard to these patients.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Regional anesthesia
Procedure: General Anesthesia — Anesthesia induction will be performed with 2.5 mg/kg propofol, 0.6 mg/kg rocuronium, and 1 mcg/kg fentanyl. Maintenance will be achieved with sevoflurane (MAC: 0.9-1.0) and remifentanil (0.05-0.2 mcg/kg/min). Remifentanil titration will be done according to basal heart rate and blood pressure.
  Tramadol (100 mg, intravenous) and dexketoprofen (50 mg, intravenous) will be administered intraoperatively as standard to these patients.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: General anesthesia

SUMMARY:
Shoulder arthroscopy is one of the most common surgical procedures performed today.It is important to perform the surgical procedure under regional anesthesia to prevent intraoperative complications due to general anesthesia.After shoulder surgery, providing adequate analgesia is necessary for both the comfort of the patient and the ability to perform the necessary post-operative rehabilitation exercises early and regularly.

Nerve blocks reduces opioid consumption in the postoperative period by providing better pain control and therefore has advantages such as fewer side effects and less risk of pulmonary and cardiac complications.

In this study; it was aimed to compare postoperative pain scores, patient satisfaction and surgeon satisfaction in patients who were operated under general anesthesia or who underwent shoulder arthroscopy while awake under regional anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* American Society of Anesthesiologists (ASA) score I-II-III
* Body Mass Index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* ASA score IV and above
* BMI below 18 or above 30 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-07-11 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | At the 0st, 1st, 2nd,4th, 12th, and 24th hours after the surgery.
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Patient satisfaction | Up to 24 hours after surgery
  Likert scale will be used to evaluate patient satisfaction (5:very satisfied, 4:satisfied, 3:undecided, 2:not satisfied, 1:very dissatisfied)
Surgeon satisfaction | Up to 24 hours after surgery
  Likert scale will be used to evaluate surgeon satisfaction (5:very satisfied, 4:satisfied, 3:undecided, 2:not satisfied, 1:very dissatisfied)
Duration of the surgery | During surgery
  For general anesthesia:
  The time from induction to extubation. For regional anesthesia: The time from the application of the block to the end of the surgery.
Intraoperatif opioid consumption | During surgery
  The amount of remifentanil used during surgery will be recorded. Remifentanil titration will be done according to basal heart rate and blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)